CLINICAL TRIAL: NCT04918498
Title: Application of Early Physical Therapy Regimens in Patients With Veno-venos Extracorporeal Membrane Oxygenation
Acronym: VV-ECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Second Affiliated Hospital of Jiaxing University (Other); Yuhang Hospital (Unknown); Changxing People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0205
Record Dates: First submitted 2021-05-31; First posted 2021-06-08 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-05

CONDITIONS: Extracorporeal Membrane Oxygenation Complication

STUDY DESIGN:
Intervention Model Description: Non-contemporaneous control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine treatment (Placebo Comparator): Review the collection of patient-related clinical data, collation of clinical data and outcome indicators
  Interventions: Behavioral: routine treatment
- Experimental group (Experimental): Implement early physiotherapy programs. The early physiotherapy program for VV-ECMO patients mainly includes the establishment of multidisciplinary teams, safety assessment, early activity physiotherapy and respiratory physiotherapy.
  Interventions: Behavioral: early physiotherapy programs

INTERVENTIONS:
Behavioral: early physiotherapy programs — establishment of multidisciplinary teams, safety assessment, early activity physiotherapy and respiratory physiotherapy
  Arms: Experimental group
Behavioral: routine treatment — provide routine nursing and rehabilitation program
  Arms: routine treatment

SUMMARY:
Promote early recovery through the application of early physiotherapy programs for VV-ECMO patients

DETAILED DESCRIPTION:
This study is intended to construct early physiotherapy programs for VV-ECMO patients, including multidisciplinary team building, safety assessment, early active physiotherapy, respiratory physiotherapy, with a view to promoting early recovery of patients, early withdrawal of ventilator-assisted ventilation, shortening ECMO auxiliary time, improving patients' exercise level and respiratory function, reducing complications, and improving the quality of near-term and long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* VV-ECMO assisted support
* lung failure (e.g. ARDS)
* age ≥18 years
* sober
* informed consent to this study

Exclusion Criteria:

* unstable blood flow mechanics
* active bleeding
* mental disorders that do not work together
* people waiting for lung transplants
* people at the end of life (e.g. advanced lung cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
VV-ECMO auxiliary time | 1 year
  the time for VV-ECMO auxiliary

CONTACTS AND LOCATIONS:
Overall Officials: Fei Zeng, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No